CLINICAL TRIAL: NCT00349492
Title: Randomized, Phase III Trial Comparing Etoposide/Cisplatin (EP) With Irinotecan/Cisplatin (IP) in Patients With Previously Untreated, Extensive Disease (ED) Small Cell Lung Cancer (SCLC)
Brief Title: A Study Comparing Etoposide/Cisplatin With Irinotecan/Cisplatin to Treat Extensive Disease Small Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinical Research Center for Solid Tumor, Korea (Other)
Responsible Party: Principal Investigator, Hyeong-Seok Lim, Dae Seog Heo, professor, Clinical Research Center for Solid Tumor, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRCST-L-0001
Record Dates: First submitted 2006-07-05; First posted 2006-07-07 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2012-03

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Extensive Disease; Chemotherapy; Randomisation
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Cisplatin

ARMS (1):
- EP (Active Comparator): etoposide + cisplatin
  Interventions: Drug: IP

INTERVENTIONS:
Drug: IP — irinotecan+cisplatin
  Other Names: irinotecan + cisplatin

SUMMARY:
This study is a randomized, multi-center clinical trial. Patients are stratified according to performance status (ECOG 0, 1 vs 2) and institution. Patients are randomized to 1 of 2 treatment arms.

Arm A: Patients receive etoposide IV on days 1, 2, 3 and cisplatin IV on day 1. Courses repeat every 3 weeks Arm B: Patients receive irinotecan IV on days 1, 8 and cisplatin IV on day 1. Coursed repeated every 3 weeks

Treatment in both arms continues for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1.5 years

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed small cell lung cancer
* Extensive disease (distant metastasis, contralateral hilar lymph node involvement, or cytologically confirmed malignant pleural effusion)
* If patients have brain metastasis with neurological symptom, they should be stabilized neurologically with prior radiotherapy or surgery for the brain metastasis (no neurologic symptom in progress and without further steroid treatment)
* No prior chemotherapy, immunotherapy, surgery or radiotherapy for small cell lung cancer (Local radiotherapy for brain or bone metastasis with symptom is permitted, in which case patients can be enrolled in this study when they have recovered from toxicity of radiotherapy)
* One or more measurable disease by RECIST criteria
* at least 18 years of age
* Performance status of 0, 1 and 2 on the Eastern Cooperative Oncology Group (ECOG) criteria
* Adequate hematologic (neutrophil count >= 1,500/uL, platelets >= 100,000/uL), hepatic (transaminase =< upper normal limit(UNL)x2.5, bilirubin level =< UNLx1.5), and renal (creatinine =< UNL) function
* Informed consent from patient which conforms to Institutional Review Board

Exclusion Criteria:

* History of cured basal cell carcinoma or cured uterine cervical malignancy except for carcinoma in situ within 5 years
* Medically uncontrolled serious heart, lung, neurological, psychological, metabolic disease
* Uncontrolled serious infection
* Enrollment in other study within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Overall survival | month

SECONDARY OUTCOMES:
Objective response rate | percent
Progression free survival | month
Safety profile | percent

CONTACTS AND LOCATIONS:
Overall Officials: Dae Seog Heo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (14):
- South Korea (14):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Yeungnam University Hospital, Daegu
  - Daegu Catholic University Hospital, Daegu
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei Cancer Center, Seoul
  - Seoul Veterans Hospital, Seoul
  - Kangnam St.Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University Medical Center, Seoul
  - Seoul Municipal Boramae Hospital, Seoul
  - St.Vincent Hospital, Suwon